CLINICAL TRIAL: NCT00543530
Title: A Noncomparative,Open, Multisite Study to Monitor the Safety and Tolerability of Efavirenz Oral Solution Given in Combination Antiretroviral Therapy (ART) in ART-naive or Experienced HIV-1 Infected Patients Age 3 to 16 Years Who Have Failed Therapy or Are Intorerant to Their Current ART Regimen
Brief Title: Pediatric Expanded Access Program-Oral Solution (0831-908)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0831-908; MK0831-908; 2007_626
Record Dates: First submitted 2007-10-05; First posted 2007-10-15 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: HIV Infections
Keywords: HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: MK0831

SUMMARY:
Monitor the safety and tolerability of efavirenz oral solution in combination with Antiretroviral Therapy for the treatment of patients age 3 to 16 years who have failed therapy or who are intolerant to their current therapy.

This is an early phase trial and some specific protocol information is in progress and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Not tolerating current ART regime laboratory status is stable
* Able to take oral liquid medications but have difficulty swallowing capsules
* Weigh at least 10 kg (22 lbs)

Exclusion Criteria:

* Has had more than 2 episodes of moderate to severe diarrhea or vomiting lasting more than 4 days within 3 months prior to taking study drug
* Have taken another investigational drug 30 days before starting this study
* Have a history of drug or alcohol abuse

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2001-03; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC